CLINICAL TRIAL: NCT02472912
Title: Single Center, Randomized, Double-Blind, 3-Way Parallel Study to Compare the Pharmacokinetics, Safety and Tolerability of BMO-2 to EU and US Sourced Humira, Administered as a Single Dose (40 mg) Subcutaneous Injection in Healthy Adults
Brief Title: Adalimumab PK Bioequivalence Study to EU and US Sourced Humira
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MYL-HEB-1001; 2014-000212-33 (EudraCT Number)
Record Dates: First submitted 2015-06-03; First posted 2015-06-16 (Estimated); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics; Adalimumab; Biosimilar Pharmaceuticals
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Single Injection of 40mg / 0.8 mL BMO-2
  Interventions: Biological: BMO-2
- Treatment B (Active Comparator): Single Injection of 40mg / 0.8 mL EU-Humira
  Interventions: Biological: EU-Humira
- Treatment C (Active Comparator): Single Injection of 40mg / 0.8 mL US-Humira
  Interventions: Biological: US-Humira

INTERVENTIONS:
Biological: BMO-2 — Volunteers randomized in Treatment A will receive a single subcutaneous injection of BMO-2 (40mg / 0.8mL).
  Other Names: Adalimumab
  Arms: Treatment A
Biological: EU-Humira — Volunteers randomized in Treatment B will receive a single subcutaneous injection of EU-Sourced Humira (40 mg / 0/8 mL)
  Other Names: Adalimumab
  Arms: Treatment B
Biological: US-Humira — Volunteers randomized in Treatment C, will receive a single subcutaneous injection of US-sourced Humira (40 mg / 0.8 mL).
  Other Names: Adalimumab
  Arms: Treatment C

SUMMARY:
Double-Blind, 3-Way Parallel Study to Compare the Pharmacokinetics, Safety and Tolerability of BMO-2 to EU and US Sourced Humira® Administered as a Single Dose (40 mg) Subcutaneous Injection in Healthy Adults.

DETAILED DESCRIPTION:
This is a single-center, randomized, double-blind, 3-way parallel study in 270 healthy adult male and female subjects. During this study, the PK bioequivalence of BMO-2, containing 40 mg adalimumab, will be compared to EU licensed Humira® (EU-Humira® ) (40 mg) and US licensed Humira® (US-Humira® ) (40 mg).

Randomization will be stratified by body weight (weight categories of 60.0-79.9 kg and 80.0-95.0 kg). After randomization, subjects will receive one of the following treatments: a single sc injection of 40 mg BMO-2, an equivalent sc injection of EU-Humira® (40 mg), or an equivalent sc injection of US-Humira® (40 mg).

Volunteers participation in the study is expected to finish with the follow-up visit, scheduled 70 days after the injection of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Weight: 60.0-95.0 kg.
* Body mass index (BMI) : 19.0-30.0 kg/m2, inclusive
* Medical history without major pathology.
* Systolic blood pressure ≤150 mmHg and diastolic blood pressure ≤90 mmHg.
* Computerized (12-lead) electrocardiogram (ECG) recording without signs of clinically relevant pathology
* Nonsmoker or light smoker
* Ability and willingness to abstain from alcohol from 48 h prior to drug administration and 48h prior to ambulatory visits, and during the stays in the clinical research center until discharge from the in-house period.
* Fertile males and females participating in heterosexual sexual relations:willingness to use adequate contraception from screening until 90 days after the follow-up visit
* Females must not lactate and must have a negative pregnancy test at screening and at admission
* Differentiation of leukocytes, platelet count, hematocrit and hemoglobin results within the reference ranges. Minor deviations considered to lack any clinical relevance by the Principal Investigator can be accepted.
* All other values for hematology and for biochemistry tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Principal Investigator.

Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* History of relevant drug and/or food allergies.
* Hypersensitivity to Humira® or its constituents.
* Known history of previous exposure to anti TNF-alpha molecules.
* Any past or concurrent medical conditions potentially increasing the subject's risks. Examples of these include medical history with evidence of clinically relevant pathology (e.g., malignancies, demyelinating disorders).
* Presence of chronic obstructive pulmonary disease (COPD). Asthma in the childhood is allowed
* Any current active infections, including localized infections, or any recent history
* Treatment with non-topical medications (including over the counter medication, and herbal remedies such as St. John's Wort extract) within 7 days prior to study drug administration, with the exception of hormonal contraceptives, multivitamins, vitamin C, food supplements and a limited amount of acetaminophen, which may be used throughout the study.
* History of active tuberculosis or presence of active or latent tuberculosis.
* Having resided or traveled in regions where tuberculosis and mycosis are endemic within 90 days before screening, or who intend to visit such a region during the period of 3 months after dosing.
* Having received live vaccines during the past 4 weeks before screening or have the intention to receive vaccination during the study.
* Participation in a drug study within 60 days or 5 half-lives of the previous drug (if known), whichever is longer, prior to drug administration
* Donation of more than 500 mL of blood within 8 weeks prior to drug administration.
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products).
* Positive urine drug screen (opiates, methadone, cocaine, amphetamines (including XTC or metamphetamines), cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants) and positive alcohol breath test.
* Positive screen on Hepatitis B surface antigen (HBsAg), anti-Hepatitis C virus antibodies (HCV), or anti-human immunodeficiency virus 1/2 antibodies (HIV).

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve (AUC) of adalimumab. | 1, 2, 3, 4, 5, 6, 7, 8, 9, 12, 15, 22, 29, 36, 43, 50, 57, 64, 71 days post subcutaneous injection.

SECONDARY OUTCOMES:
Frequency of Adverse Events | Up to 71 days.
Safey variable - Tolerability (injection site reactions) | Predose and 1, 2, 3, 7, 9, 36, and 71 days post subcutaneous injection.
  Tolerability assessments as measured by injection site reactions
Safety variable - immunogenicity (Presence of anti-adalimumab antibodies) | Day 1 (pre-dose) and Day 9, 29, and 71 days post subcutaneous injection.
  Presence of anti-adalimumab antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Principal Investigator — SGS Belgium NV; Fausto Berti, Study Director — Mylan GmbH
Locations (1):
- SGS Belgium NV, Antwerp, Belgium